CLINICAL TRIAL: NCT00852618
Title: Intensive Viral Dynamics Substudy of A5248
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: A5249s; 10618 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Treatment Naive
Keywords: HIV Integrase Inhibitors; HIV Nucleoside Reverse Transcriptase Inhibitors; Treatment Naive; Viral Load
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be collected throughout the study

GROUPS / COHORTS (2):
- A: Participants undergoing treatment with raltegravir (RAL) in the main study
- B: Participants undergoing treatment with emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) in the main study

SUMMARY:
The HIV integrase inhibitor, raltegravir (RAL), which was recently approved by the FDA, has been shown in several trials to be highly effective. The main study will estimate the viral load decay rate in treatment-naive HIV-infected participants receiving RAL and emtricitabine/tenofovir disoproxil fumarate (FTC/TDF).

This substudy of A5248 will similarly examine the characteristics of decrease in viral load but will focus on estimating the time at which first-phase viral decay starts, following initiation of the study drugs.

DETAILED DESCRIPTION:
Recent data suggest that early virologic response to HIV interventions may be predictive of long-term virologic outcomes. Defining early decay in viral load through carefully performed studies of viral dynamics may be a useful tool for assessing the likely outcome of long-term treatment. It may also be a useful screening tool to define which combinations should be studied further. In the main study, the viral load decay rate will be estimated in HIV-infected, treatment-naive participants receiving RAL and FTC/TDF.

The A5248 study will last approximately 72 weeks. All participants will take RAL and FTC/TDF for 72 weeks. RAL will be provided by the study. FTC/TDF will not be provided.

A5248 will consist of 16 study visits. These visits will occur at study entry; Days 2, 7, 10, 14, 21, 28, and 56, and Weeks 12, 16, 20, 24, 36, 48, 60, and 72. Blood collection and pharmacokinetic studies will occur at all study visits. Self-reported adherence assessments will be submitted at each visit. A targeted physical exam will occur at most visits. Liver function tests and urine collection will occur at select visits. Pregnancy tests will occur whenever pregnancy is suspected.

This substudy will enroll 10 participants from A5248. It is critical that substudy participants take their medications as directed to ensure accurate trial results. Any participant who discontinues study treatment will also be removed from the substudy and replaced. Participants will be asked about medication holds and adherence.

No medications will be provided by the substudy. Study treatment will be provided and administered as per the main study, A5248. After participants begin study medications, samples will be collected for the substudy. Participants will be required to stay overnight and in the hospital from Day 0 until Day 2. The morning study medication dose will be administered in the clinic on Days, 2, 3, 4, and 7.

Medication diaries will be provided for participants on Day 2. Participants will be instructed to record the times they take their study medications through Day 7 of the study. Participants are required to bring these diaries to their study visits on Days 3, 4, and 7 for review.

Participants may discontinue their enrollment in this substudy and still remain in the main study, A5248. Participants may not discontinue their involvement in A5248 and remain in the substudy.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in A5248
* Willing and able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected participants currently enrolled in study A5248
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-05; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Time at which first-phase viral decay begins | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Andrade, MD, MPH, Study Chair — Johns Hopkins University
Locations (6):
- United States (6):
  - University of Colorado Hospital CRS, Aurora, Colorado
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Trillium Health ACTG CRS, Rochester, New York
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee